CLINICAL TRIAL: NCT04149691
Title: A Phase I, Open-label, Multicentre, Dose Escalation Study to Assess Safety, Tolerability and Pharmacokinetics of Oral CPL304110, in Adult Subjects With Advanced Solid Malignancies
Brief Title: Safety, Tolerability and Pharmacokinetics of Oral CPL304110, in Adult Subjects With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01FGFR2018
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Bladder Cancer; Squamous Non-small Cell Lung Cancer; Cholangiocarcinoma; Sarcoma; Endometrial Cancer; Other Solid Tumours
Keywords: FGFR; kinase inhibitor; advanced solid tumors; carcinoma; neoplasms; gastric cancer; bladder cancer; squamous non-small cell lung cancer; squamous immunophenotype
MeSH Terms: conditions — Stomach Neoplasms; Urinary Bladder Neoplasms; Cholangiocarcinoma; Sarcoma; Endometrial Neoplasms; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPL304110 (Experimental): CPL304110 will be administered once daily to adults with advanced solid malignancies in 28-day cycles.
  Interventions: Drug: CPL304110

INTERVENTIONS:
Drug: CPL304110 — CPL304110 is to be administered orally as hard gelatine capsules once daily in 28-day cycles.
  Other Names: PG19

SUMMARY:
The purpose of the study is to determine to evaluate safety and tolerability of CPL304110 when administered once daily to adults with advanced solid malignancies.

DETAILED DESCRIPTION:
01FGFR2018 is an Open-label, Multicentre, Dose Escalation Study to Assess Safety, Tolerability and Pharmacokinetics of Oral CPL304110, in Adult Subjects with Advanced Solid Malignancies. The study consists of 3 parts: initial dose escalation (Part 1 - without FGFR, fibroblast growth factor receptor, molecular aberrations), dose escalation (Part 2 - with FGFR molecular aberrations) and dose extension (Part 3 - with FGFR molecular aberrations).

ELIGIBILITY:
Inclusion Criteria:

* Patient or legal guardian, if permitted by local regulatory authorities, provides informed consent to participate in the study must be performed before any procedure's protocol related
* age of ≥25 years old
* Performance Score ≥70 in accordance with the Karnofsky Performance Score (KPS),
* life expectancy period of at least 3 months on the screening day,
* Have measurable disease according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
* subject (or his/her partner) of childbearing potential willingness to use acceptable forms of contraception
* adequate blood, liver, renal and urine parameters
* phosphate levels within normal range
* HIV, HCV (hepatitis C virus) and HBV negative (hepatitis B virus),
* adequate cardiac function

Inclusion Criteria Specific for parts:

Part 1

* Patients with histologically confirmed advanced gastric cancer, bladder cancer, squamous lung cancer or non-small cell lung cancer with squamous immunophenotype, cholangiocarcinoma, sarcoma or endometrial cancer, be refractory to prior therapies and without effective further treatment options.

Part 2 and 3

* Patients with histologically confirmed advanced gastric cancer, bladder cancer, squamous lung cancer or non-small cell lung cancer with squamous immunophenotype, be refractory to prior therapies and without effective further treatment options.
* Subject's archival formalin-fixed paraffin-embedded (FFPE) tumour sample available for molecular alteration diagnostics, and/or a possibility to collect a new biopsy.
* Present molecular alteration within FGFR 1, 2 or 3

Exclusion Criteria:

* Any other current malignancy or malignancy diagnosed within the past five (5) years.
* Active brain metastases or leptomeningeal metastases.
* concurrent anticancer treatment within 28 days before the start of trial treatment; major surgery within 28 days before the start of trial treatment); use of blood transfusion within 7 days before the start of trial treatment,
* prior therapy with an agent directed to another FGFR inhibitor,
* pregnancy and/or breastfeeding,
* phosphate levels above the upper limit of normal,
* ectopic calcification/mineralization,
* endocrine alteration related to calcium/phosphate homeostasis e.g. parathyroid disorders, history of parathyroidectomy,
* concomitant therapies increasing calcium/phosphate serum levels,
* inability to take oral medicines,
* corneal disorder and/or keratopathy,
* persisting toxicity related to prior therapy Grade > 1 CTCAE v5.0, except polyneuropathy and alopecia,
* clinically significant (i.e., active) cardiovascular disease. History of abdominal fistula, bowel obstruction (Grade IV), gastrointestinal perforation, intra-abdominal abscess within 6 months of enrollment. Other significant diseases, which, in the opinion of the investigator, might impair the subject's tolerance of trial treatment.
* Receipt of any organ transplantation including allogeneic stem-cell transplantation.

Exclusion Criteria Specific for parts:

Part 2 and 3

* No FFPE tumour sample available to conduct FGFR alteration eligibility tests and no biopsy option.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | First cycle of 28 days
  Maximum tolerated dose (MTD) of CPL304110 when administered orally once daily to adults with advanced solid malignancies. The MTD is the highest dose associated with the occurrence of dose-limiting toxicities (DLTs) in <33% of patients.
Safety profile | First cycle of 28 days
  Overall safety profile of CPL304110, as assessed by the type, frequency, severity, timing, and relationship to study drug of any adverse events (AEs), serious adverse events (SAEs), and changes in vital signs, ECGs, and safety laboratory test.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) determined on the base of the MTD. | Approximately up to 12 months
  The RP2D will be determined after review and discussion of the pharmacokinetics (PK) profile, type and severity of drug related toxicity and clinical suitability for long-term administration.
ORR, objective rate response | Approximately up to 12 months
  ORR, objective rate response defined as the rate of confirmed complete response (CR) or partial response (PR) by RECIST 1.1.
Maximum plasma concentration (Cmax) | up to 24 hours after CPL304110 administration
  Cmax defines the maximum concentration of the product in plasma during observation period.
Time to maximum plasma concentration (tmax) | up to 24 hours after CPL304110 administration
  tmax defines Time to reach maximum plasma concentration
Area under the plasma concentration versus time curve (AUC) from 0 up to the time of last quantifiable concentration (AUC0-t) | up to the time of last quantifiable concentration after CPL304110 administration
  AUC(0-t) defines the area under the curve of plasma concentration vs time, from time point zero up to the time of last quantifiable concentration
Area under the plasma concentration versus time curve AUC from 0 to infinity (AUC0-inf) | up to 24 hours after CPL304110 administration
  AUC0-inf defines the area under the curve of plasma concentration vs time, from time point zero extrapolated to infinity
Terminal half-life (t½) | up to 24 hours after CPL304110 administration
  Plasma elimination half-life
Kel: Terminal elimination rate constant | up to 24 hours after CPL304110 administration
  Terminal elimination rate constant

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk
  - BioResearch Group sp. z o.o., Nadarzyn
  - SP ZOZ MSWiA z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Klinika Onkologii, Europejskie Centrum Zdrowia, Otwock
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie, Warsaw
  - Instytut Gruźlicy i Chorób Płuc, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamani A, Zdzalik-Bielecka D, Lipner J, Stanczak A, Piorkowska N, Stanczak PS, Olejkowska P, Hucz-Kalitowska J, Magdycz M, Dzwonek K, Dubiel K, Lamparska-Przybysz M, Popiel D, Pieczykolan J, Wieczorek M. Discovery and optimization of novel pyrazole-benzimidazole CPL304110, as a potent and selective inhibitor of fibroblast growth factor receptors FGFR (1-3). Eur J Med Chem. 2021 Jan 15;210:112990. doi: 10.1016/j.ejmech.2020.112990. Epub 2020 Nov 7. PMID 33199155